CLINICAL TRIAL: NCT06113406
Title: Evaluation of Virtual Reality in Hazmat Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetaMedia Training International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R43ES034218 (NIH)
Record Dates: First submitted 2023-06-13; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: No Disease or Condition is Being Studied; Evaluating a Brief Intervention; Does Virtual Reality Aid in Hazmat Training

STUDY DESIGN:
Intervention Model Description: An experimental and a pretest-posttest control group design method were applied in this regard.
Who Masked: Outcomes Assessor
Masking Description: The person who will make the statistical analysis does not know which group the participants in our study belong to and does not know the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classroom Training (Active Comparator): The active control group is given traditional hazmat response training which is already part of their curriculum. For the traditional training group the session is given in the classroom for 45 minutes and the training session is ended.
  Interventions: Behavioral: Classroom Training
- Virtual Reality Training (Experimental): After the traditional training has ended, the experimental group will receive the additional VR scenario, online educational content and question and answer session. For the VR training group, the participant is asked to perform the analyze, plan, implement, and evaluation steps individually. After the training is completed the session is closed.
  Interventions: Behavioral: Virtual Reality Training

INTERVENTIONS:
Behavioral: Classroom Training — Active Comparator
  Arms: Classroom Training
Behavioral: Virtual Reality Training — Experimental
  Arms: Virtual Reality Training

SUMMARY:
Type of study: Two-group comparison.

Main question it aims to answer:

Does the use of virtual reality emergency scenarios provide a practical and effective tool to supplement traditional instructor-led training for first responder trainees?

A. For the traditional hazmat response training group; Traditional training will be held in the classroom environment for 45 minutes in the form of a lecture, then the training session will be terminated.

B. For VR hazmat response training group; After the traditional classroom session has ended, the participants will complete the additional VR training scenario, online content, and question-answer session. Once completed the session will be closed.

ELIGIBILITY:
Inclusion Criteria:

* currently enrolled in a hazmat training course

Exclusion Criteria:

* under the age of 18 or over the age of 65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Keywords identified on questionnaire | day 1
  Participants will receive a score of zero to ten based on the number of keywords they identified. Each correct key word identified is worth 1 point. Minimum 0, maximum 10 points can be scored. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- MetaMedia Training International, Frederick, Maryland, United States

IPD SHARING:
Plan to Share IPD: No